Title:

The Effects of Vitamin D Supplementation on Glycemic Control in Children with Type 1 Diabetes

Mellitus in Gaza Strip, A Randomized Controlled Trial.

**Authors:** 

Heba AbdAllah Al Sarraj<sup>1</sup>, Ashraf Jaber Shaqaliah<sup>1</sup>, Heba Mohammed Arafat<sup>2</sup>, Ohood

Mohammed Shamallakh<sup>3</sup>, and Kholoud Mohammed Shamallakh<sup>3</sup>.

**Affiliations:** 

<sup>1</sup> Department of Laboratory Medicine, Al Azhar University-Gaza, Gaza Strip, Palestine;

hebasarraj24@gmail.com; ashshaq@yahoo.com.

<sup>2</sup> Department of Chemical Pathology, School of Medical Sciences, Health Campus, Universiti

Sains Malaysia, Kubang Kerian, Kelantan, Malaysia; <a href="hebaarafat4@usm.my">hebaarafat4@usm.my</a>.

<sup>3</sup> Department of a Medical Laboratory Sciences, Faculty of Health Sciences, Islamic University of

Gaza, Gaza City, Palestine; oho.od@hotmail.com; loody89@windowslive.com.

**Running title:** 

Vitamin D Supplementation and Glycemic Control Improvement among Type 1 Diabetic

Children

**Corresponding Author:** 

Heba Mohammed Arafat

Department of Chemical Pathology, School of Medical Sciences, Health Campus, Universiti Sains

Malaysia, Kubang Kerian, Kelantan, Malaysia.

Email: hebaarafat4@usm.my.

Phone Number: +972599575745.

**Document Date**: November 14, 2021

## Statistical analysis

- Statistical Package for the Social Science (SPSS, version 22) was used for data processing and analysis.
- Description of variables was presented as follows:
- Data were normally distributed, as determined using Kolmogorox-Smirnov test.
- Description of quantitative variables were presented as the following: Normally distributed data were expressed as mean  $\pm$  SD.
- Description of qualitative variables was in the form of numbers (No.) and percent (%).
- Comparison between quantitative variables was carried out by student T-test of two independent samples. Results were expressed in the form of P-values.
- Comparison between qualitative variables was carried out by Chi-Square test (χ²).
  Fisher exact test was used instead of Chi- square test when one expected cell or more were ≤ 5.
- Binary correlation was carried out by Spearman correlation test. Results were expressed in the form of correlation coefficient (R) and P-values. The following points are the accepted guidelines for interpreting the correlation coefficient:
  - 0 indicates no linear relationship.
  - +1 indicates a perfect positive linear relationship: as one variable increases in its values, the other variable also increases in its values via an exact linear rule.

## Sample size calculation

To calculate the sample size two mean formula was used as follow

$$n = \frac{2\sigma^2}{\Delta^2} \left( z_{\alpha/2} + z_{\beta} \right)^2$$

 $\sigma = 67.8$  Bilateral large drusen

 $\Delta = 50$  (expected improvement in the Bilateral large drusen after intervention

$$Z(\alpha/2) = 1.96$$
 for  $\alpha = 0.05$  (two-tailed)

 $z_{-}(\beta) = 0.84 \text{ for } 80\% \text{ power}$ 

$$n = \frac{2(67.8)^2}{(50)^2} (1.96 + 0.84)^2$$

$$n = 28.8 = 29$$

Total number of cases = 29 + non response rate 20%

n = 29 + 6 = 35 cases in each group